CLINICAL TRIAL: NCT05523024
Title: Effect of Probiotics or Berberine Supplementation on Hepatic Steatosis Markers, Cardiometabolic and Microbiotic Profile in NAFL - A Randomized Double- Blind Clinical Study.
Brief Title: Effect of Probiotics or Berberine in Hepatic Steatosis Markers, Cardiometabolic and Microbiotic Profile in NAFL.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 491/20;
Record Dates: First submitted 2022-04-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Non Alcoholic Fatty Liver; Obesity
Keywords: NAFL; obesity; probiotics; berberine; microbiota;
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Probiotics; Berberine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotic (Active Comparator): Individuals receive Probiotics (9 strains: B. bifidum W23, B. lactis W51, B. lactis W52, L. acidophilus W37, L. brevis W63, L. casei W56, L. salivarius W24, Lactococcus lactis W19, and Lactococcus lactis W58) in dose: 1x109 colony forming units (CFU), daily, for 12 weeks.
  Intervention: Dietary Supplement: Probiotic
  Interventions: Dietary Supplement: Probiotic
- Berberine (Active Comparator): Individuals receive Berberine (Berberine hydrochloride 97% extract of Berberis aristata) in dose: 1500 mg/day, for 12 weeks.
  Intervention: Dietary Supplement: Berberine
  Interventions: Dietary Supplement: Berberine
- Placebo (Placebo Comparator): Individuals receive placebo daily, for 3 months. Intervention: Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo
- Probiotics and Berberine (Active Comparator): Individuals receive: Probiotics (9 strains: B. bifidum W23, B. lactis W51, B. lactis W52, L. acidophilus W37, L. brevis W63, L. casei W56, L. salivarius W24, Lactococcus lactis W19, and Lactococcus lactis W58) in dose: 1x109 colony forming units (CFU), daily and Berberine (Berberine hydrochloride 97% extract of Berberis aristata) in dose: 1500 mg/day, for 12 weeks.
  Intervention: Dietary Supplement: Probiotic and Berberine
  Interventions: Dietary Supplement: Probiotc and Berberine

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic group will receive one capsule of the probiotic mixture (dose:1x109 colony forming units (CFU) per day in one dose (before breakfast). The PRO preparation will contain the following bacterial strains: 50% Lactococcus lactis Rosell® - 1058, 25% Lactobacillus casei Rosell® - 215, 12,5% Lactobacillus helveticus Rosell® - 52, 12,5% Bifidobacterium bifidum Rosell® - 71). Probiotics will be administered orally.
  Arms: Probiotic
Dietary Supplement: Berberine — The berberine group will receive 1500 mg of Berberine (Berberine hydrochloride 97% extract of Berberis aristata) per day in 3 doses. Berberine will be administered orally, before breakfast, dinner, and before supper.
  Arms: Berberine
Dietary Supplement: Placebo — The placebo group will receive a placebo. Placebo will contain only the excipients and will be administered orally for 24 weeks. Placebo in no way: color, taste, smell, form of taking, the dosage will not differ from the preparations tested. However, it will not contain probiotcs or berberine. Placebo will be orally administered three times a day: before breakfast, dinner, and supper (6.00-7.00 p.m.). To meet the GCP conditions, subjects from all groups will receive the same number of capsules (six) per day.
  Arms: Placebo
Dietary Supplement: Probiotc and Berberine — Probiotics and Berberine groupwill receive both: a probiotics mixture (as in PRO group: 1x109 CFU/day; in one dose) and 1500 mg/day of Berberine (Berberine hydrochloride 97% extract of Berberis aristata; in 3 doses). Probiotcs and berberine will be administered orally before breakfast, before dinner, and before supper.
  Arms: Probiotics and Berberine

SUMMARY:
Effect of oral selected Probiotics (PRO) and/or Berberine (BBR) supplementation on hepatic steatosis markers, cardiometabolic profile, and gut microbiota profile in the non-alcoholic fatty liver (NAFL) - a randomized double-blind clinical study.

DETAILED DESCRIPTION:
Probiotics (PRO) and bioactive natural substances such as Berberine (BBR) can improve metabolic parameters in patients with obesity and metabolic disorders. In addition, they significantly affect the composition and function of gut microbiota (GM) and support anti-inflammation and antioxidant defense. These data have become the starting point for the proposed multidirectional approach, aimed at assessing the effect of PRO and/or BBR supplementation on:

* hepatic-related outcomes,
* changes in anthropometric measurements (body mass, BMI, body mass composition and fat mass % content),
* cardiometabolic profile (e.g. blood pressure, noninvasive markers of endothelial function, cardiometabolic biochemical parameters)
* microbiotic profile (gut microbiota composition, endotoxemia)
* the content of the minerals, in overweight/obese patients with nonalcoholic fatty liver (NAFL).

ELIGIBILITY:
Inclusion Criteria:

* age 40 to 60 years;
* women ≥1 year since last menstruation;
* body mass index (BMI): 27.0 kg/m2 to 34.9 kg/m2;
* abdominal obesity-related waist circumference > 80 cm (women) and >94 cm (men) (in accordance to International Diabetes Federation);
* stable body weight in the 3 months prior to the trial (permissible deviation is ± 3 kg);
* NAFL - diagnosed based on USG in accordance with PGE-NAFLD recommendation

Exclusion Criteria:

* history of following alternative diets within 3 months before the study;
* history of use of any dietary supplements in the 3 months before the study;
* history of intake of antibiotics, probiotics, prebiotics within 3 months before the study;
* secondary form of obesity, pharmacological treatment for obesity (in the 3 months before the study), history of bariatric surgery;
* another liver diseases: high risk of NASH (assessed on the FIB-4, according to the PGE-NAFLD recommendation), autoimmune hepatitis, hepatitis B and C, toxic hepatitis, cirrhosis, Wilson's disease, hemochromatosis;
* other gastrointestinal disorders, especially: IBD, celiac disease, gastritis and duodenitis, pancreatic disorders, gastrointestinal symptoms suggestive of IBS;
* clinically significant acute inflammatory process (elevated hsCRP);
* abnormal kidney function (GFR <60mL/min/1,73m2);
* T2D;
* dyslipidemia or hypertension - requiring the introduction and/or change of pharmacological treatment in the 6 months before the trial or during intervention;
* pump inhibitors, anticoagulants, drugs causing metabolic alteration, e.g., SFAs (second-generation antipsychotics);
* diseases requiring nutritional requirement and chronic supplementation;
* alcohol (>30g/d for men and >20g/d for women), nicotine or drug abuse;
* mental disorders, including eating disorders;
* cancer, autoimmune diseases;
* any other condition which may influence on final results of the study or pose a risk for subjects health.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Fibrosis-4 (FIB-4) - Index for Liver Fibrosis. | At the baseline and 12 weeks of treatment
  FIB-4 will be estimated using a medical calculator (based on parameters as: age, ALT, AST, and platelet count).
Changes in HSI - Hepatic Steatosis Index. | At the baseline and 12 weeks of treatment
  HSI will be estimated using a medical calculator (based on parameters as: gender, ALT, AST, BMI, and type 2 diabetes).
Changes in NAFLD-LFS (liver fat score). | At the baseline and 12 weeks of treatment
  NAFLD-LFS will be estimated using a medical calculator (based on serum aspartate transaminase/alanine transaminase (AST/ALT) ratio, fasting serum aspartate transaminase (AST) level, fasting serum insulin level, presence of metabolic syndrome and diabetes mellitus).

SECONDARY OUTCOMES:
Changes in blood pressure. | At the baseline and 12 weeks of treatment
  Resting seated BP (both systolic and diastolic) will be measured using a brachial cuff (Omron Healthcare, Kyoto, Japan) three times at 2-min intervals, and the average value will be calculated.
Changes in weight. | At the baseline and 12 weeks of treatment
  Weight will be measured in light clothing and without metal objects (i.e., belt, jewelry). Weight will be measured to the nearest 0.1 kg.
Changes in waist circumference, hip circumference. | At the baseline and 12 weeks of treatment
  WC will be measured between the iliac crest and the lower rib at the end of a normal expiration, and HC will be measured around the widest portion of the buttocks. Both HC and WC will be measured using stretch-resistant medical tape (Seco) to the nearest 0.5 cm. The measurement of WC and HC will be performed according to the World Health Organization (WHO) protocol.
Changes in waist to hip ratio. | At the baseline and 12 weeks of treatment
  WHR will be calculated as WC to HC quotient.
Changes in BMI. | At the baseline and 12 weeks of treatment
  BMI will be calculated according to the formula: BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meters squared.
Changes in fat mass content in the body. | At the baseline and 12 weeks of treatment
  The fat mass content [in kg] in the body will be estimated using BIA methods (InBody 270 and Bioscan 920-2),
Changes in pulse wave velocity (PWV). | At the baseline and 12 weeks of treatment
  The pulse wave velocity (PWV) will be measured using the SphygmoCor Px (Atcor Medical Blood Pressure Analysis System, Sydney, Australia) in a temperature-controlled room before making anthropometric measurements and blood collection.
Changes in pulse wave analysis (PWA). | At the baseline and 12 weeks of treatment
  The pulse wave analysis (PWA)will be measured using the SphygmoCor Px (Atcor Medical Blood Pressure Analysis System, Sydney, Australia) in a temperature-controlled room before making anthropometric measurements and blood collection.
Gut (taxonomic and functional) microbiota analysis in stool. | At the baseline and 12 weeks of treatment
  Analyzed by the NGS method.
Short-chain fatty acids (SCFAs) concentration in stool. | At the baseline and 12 weeks of treatment
  Analyzed using gas chromatography (Agilent Technologies 1260 A GC system with a flame ionization detector (FID))
Measurement of hair minerals (Fe, Mg, Ca, Cu, Zn) concentration. | At the baseline and 12 weeks of treatment
  Performed using atomic absorption spectrometry (Atomic Absorption Spectrophotometer ZA3000, Hitachi, Tokyo, Japan)
Changes in ALT, AST, GGT | At the baseline and 12 weeks of treatment
  The ALT, AST, GGT will be measured using standard methods.
Changes in non-esterified free fatty acids. | At the baseline and 12 weeks of treatment
  The NEFA will be measured using standard methods.
Changes in lipids profile (TC, HDL, TG). | At the baseline and 12 weeks of treatment
  The TC, HDL, TG will be measured using standard methods.
Changes in low-density lipoprotein (LDL). | At the baseline and 12 weeks of treatment
  The low-density lipoprotein cholesterol (LDL) will be calculated according to the Friedwald equation.
Changes in fasting glucose level. | At the baseline and 12 weeks of treatment
  The fasting glucose level will be measured using standard methods.
Changes in fasting insulin level. | At the baseline and 12 weeks of treatment
  The ELISA will be used in the estimation.
Changes in insulin resistance index (HOMA-IR) | At the baseline and 12 weeks of treatment
  The HOMA-IR will be calculated according to formula:
  HOMA-IR = (insulin * glucose) / 22.5 for the glucose concentration in mmol/L, or: HOMA-IR = (insulin * glucose ) / 405 for glycemia in mg/dL. In both cases, the insulin is in mU/L.
Changes in parameter of liver damage: cytokeratin 18. | At the baseline and 12 weeks of treatment
  The ELISA will be used in the estimation cytokeratin 18 (ccK18).
Changes in parameter of liver damage: Glutathione S-transferase (GST). | At the baseline and 12 weeks of treatment
  The ELISA will be used in the estimation GST.
Changes in parameter of liver damage: collagen IV. | At the baseline and 12 weeks of treatment
  The ELISA will be used in the estimation collagen IV.
Changes in parameter of liver damage: hyaluronic acid. | At the baseline and 12 weeks of treatment
  The ELISA will be used in the estimation hyaluronic acid.
Changes in hsCRP. | At the baseline and 12 weeks of treatment
  The hsCRP will be measured using ELISA.
Changes in pentraxin 3. | At the baseline and 12 weeks of treatment
  The pentraxin 3 (PTX3) will be measured using ELISA.
Gut barrier integrity parameter: calprotectin. | At the baseline and 12 weeks of treatment
  The ELISA, will be used in the estimation.
Gut barrier integrity parameters: liver fatty acid-binding protein (L-FABP), intestinal fatty acid-binding protein (I-FABP). | At the baseline and 12 weeks of treatment
  The ELISA, will be used in the estimation.
Gut barrier integrity parameters: lipopolysaccharide (LPS). | At the baseline and 12 weeks of treatment
  The ELISA, will be used in the estimation.
Cardiometabolic risk. | At the baseline and 12 weeks of treatment
  Cardiometabolic risk will be estimated at baseline and after 3 months of treatment using the SCORE scale. SCORE scale summarize 5 risk factors (sex, age, systolic blood pressure, total cholesterol and smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Bogdański, Professor, Principal Investigator — Poznan University of Medical Sciences, Poznan, Poland
Locations (1):
- 2 Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics, Poznań University of Medical Sciences,, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No